CLINICAL TRIAL: NCT00002560
Title: PHASE II TRIAL OF MONOCLONAL ANTIBODY 3F8 AND GRANULOCYTE-MACROPHAGE COLONY-STIMULATING FACTOR (GM-CSF) FOR NEUROBLASTOMA
Brief Title: Monoclonal Antibody Therapy Plus Sargramostin in Treating Patients With Advanced Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 94-018; CDR0000063466 (Registry Identifier: PDQ (Physician Data Query)); NCI-V94-0416
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody; sargramostim

INTERVENTIONS:
Biological: monoclonal antibody 3F8
Biological: sargramostim

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining colony-stimulating factors, such as sargramostim, with monoclonal antibodies may be an effective treatment for advanced neuroblastoma.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody 3F8 plus sargramostim in treating patients who have advanced neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the antitumor effects of monoclonal antibody 3F8/sargramostim (3F8/GM-CSF) in patients with advanced neuroblastoma.
* Assess the biological effects of 3F8/GM-CSF in these patients.

OUTLINE: Patients receive monoclonal antibody 3F8 IV over 1.5 hours on days 0-4 and 7-11 and sargramostim (GM-CSF) IV over 2 hours on days -5 to 11. Treatment is repeated every 4 weeks for up to 4 courses in the absence of progressive disease, HAMA response, or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 11-40 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Neuroblastoma diagnosed by INSS criteria, i.e., either:

  * Histologic proof of disease OR
  * Tumor clumps in bone marrow plus elevated catecholamine levels
* Relapsed disease with poor long-term prognosis as indicated by at least one of the following:

  * N-myc amplification in tumor cells
  * Diploid chromosomal content in tumor cells
  * Distant skeletal metastases
  * Unresectable primary tumor crossing the midline
  * Bone marrow with greater than 10% tumor cells
* Documentation of measurable progressive disease or biopsy- proven stable disease at least 4 weeks after prior systemic therapy required
* No rapidly progressive disease
* Poor risk neuroblastoma (but without measurable disease) not eligible for other neuroblastoma protocols

PATIENT CHARACTERISTICS:

Age:

* 2 to 21

Performance status:

* Not specified

Life expectancy:

* Greater than 8 weeks

Hematologic:

* Not specified

Hepatic:

* No grade 3/4 toxicity
* LDH no greater than 1.5 times upper limit of normal

Renal:

* Creatinine clearance at least 60 mL/min
* No grade 3/4 toxicity

Cardiovascular:

* No grade 3/4 toxicity

Pulmonary:

* No grade 3/4 toxicity

Other:

* No grade 3/4 neurologic, gastrointestinal, or other organ toxicity except grade 3 hearing deficit
* No active life threatening infections
* No human antimouse antibody (HAMA) greater than 1,000 ELISA units/mL
* No allergy to mouse proteins
* No pain requiring opiates

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Standard chemotherapy to which disease is resistant or myeloablative therapy followed by disease recurrence required

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 1994-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian H. Kushner, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States